CLINICAL TRIAL: NCT00604565
Title: A Prospective, Randomized, Open-label, Multi-center, Controlled Clinical Trial of the Safety and Efficacy of Physiological Iron Maintenance in End Stage Renal Disease (ESRD) Subjects by Delivery of Soluble Ferric Pyrophosphate (SFP) Via Hemodialysate
Brief Title: Delivery of Soluble Ferric Pyrophosphate (SFP) Via the Dialysate to Maintain Iron Balance in Hemodialysis Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: major planned changes to study design
Sponsor: Charles Drew University of Medicine and Science (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Rockwell Medical Technologies, Inc. (Industry)
Responsible Party: Principal Investigator, Ajay Gupta, Ajay Gupta, MD, Charles Drew University of Medicine and Science
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: SFP-NIH-01; NIH-FP-01
Record Dates: First submitted 2008-01-17; First posted 2008-01-30 (Estimated); Results first posted 2015-08-31 (Estimated); Last update posted 2015-08-31 (Estimated); Status verified 2015-08

CONDITIONS: End Stage Renal Disease (ESRD)
Keywords: Hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- SFP dialysate (Experimental): dialysate with added soluble ferric pyrophosphate (SFP)
  Interventions: Drug: soluble ferric pyrophosphate (SFP)
- standard dialysate (Placebo Comparator): standard dialysate without soluble ferric pyrophosphate (SFP)
  Interventions: Other: placebo

INTERVENTIONS:
Drug: soluble ferric pyrophosphate (SFP) — Subjects will be randomized to undergo dialysis with either Fe-HD (dialysate containing SFP) The experimental concentrate containing SFP (Fe-HD)has 95mg of SFP per gallon, or 10.9 mg total iron per gallon (96 µg of SFP per dL or 11 µg of total iron per dL).
  Control concentrate lacking SFP (C-HD) does not contain SFP (total iron = 0)
  Arms: SFP dialysate
Other: placebo — Subjects will be randomized to undergo dialysis with C-HD (conventional dialysate lacking SFP)
  Arms: standard dialysate

SUMMARY:
In maintenance hemodialysis patients, regular administration of parenteral iron by addition of soluble ferric pyrophosphate (SFP) to the dialysate, when compared to conventional dialysate, is effective in preventing the development of iron deficiency, thereby maintaining hemoglobin level; is clinically safe and does not lead to oxidative stress or inflammation.

ELIGIBILITY:
Inclusion Criteria:Subjects with end stage renal disease undergoing maintenance hemodialysis three times a week.

* Subjects who have required IV iron at any time in the 2 months preceding enrollment.

Exclusion Criteria:

* Subjects with absolute iron deficiency at the time of enrollment In hemodialysis subjects "absolute iron deficiency"
* Subjects with a current malignancy involving sites other than skin.
* Subjects with a history of drug or alcohol abuse within the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2008-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Gupta, MD, Principal Investigator — Rockwell Medical Technologies, Inc.
Locations (2):
- United States (2):
  - RAI, Los Angeles, California
  - University of Louisville Kidney Disease Program, Louisville, Kentucky

RESULTS

PARTICIPANT FLOW:
Groups:
- SFP Dialysate: dialysate with added soluble ferric pyrophosphate (SFP)
  soluble ferric pyrophosphate (SFP): Subjects will be randomized to undergo dialysis with Fe-HD (dialysate containing SFP) The experimental concentrate containing SFP (Fe-HD)has 95mg of SFP per gallon, or 10.9 mg total iron per gallon (96 µg of SFP per dL or 11 µg of total iron per dL).
Period: Overall Study
Arm/Group | SFP Dialysate | Standard Dialysate
Started | 4 | 7
Completed | 4 | 4
Not Completed | 0 | 3
Not completed — Study terminated | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SFP Dialysate | Standard Dialysate | Total
Number analyzed (Participants) | 4 | 7 | 11
Age, Continuous [Mean (Full Range); unit: years] | 51.5 [39 to 67] | 55.4 [41 to 65] | 54.0 [39 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 1 | 5 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 5 | 6
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 4 | 7 | 11

OUTCOME MEASURES:

1. Primary Outcome: TOTAL NUMBER OF SUBJECTS WITH ADVERSE EVENTS
Description: Incidence and seriousness of adverse events will be captured from date of randomization until study participation completion (up to 36 weeks). For the Primary Outcome Measure, total number of subjects affected are listed only. The details of the types of events that took place are reported in the Adverse Events section.
Time Frame: 36 weeks
Population: All subjects were included in the Safety Analysis population.
Measure: Number; unit: participants
Arm/Group | SFP Dialysate | Standard Dialysate
Number analyzed (Participants) | 4 | 7
participants
  Number of Subjects Who Experienced Serious AE | 0 | 1
  Number of Subjects Who Experienced Non-serious AE | 4 | 7

2. Primary Outcome: TOTAL NUMBER OF ADVERSE EVENTS
Description: Incidence and seriousness of adverse events will be captured from date of randomization until study participation completion (up to 36 weeks). For the Primary Outcome Measure, total number of events are listed only. The details of the types of events that took place are reported in the Adverse Events section.
Time Frame: 36 weeks
Population: All subjects were included in the Safety Analysis population.
Measure: Number; unit: events
Arm/Group | SFP Dialysate | Standard Dialysate
Number analyzed (Participants) | 4 | 7
events
  Total Number of Serious Adverse Events (SAEs) | 0 | 1
  Total Number of Non-Serious Adverse Events | 66 | 115

ADVERSE EVENTS:
Arm/Group | SFP Dialysate | Standard Dialysate
Serious Adverse Events (participants affected / at risk) | 0/4 | 1/7
Other Adverse Events (participants affected / at risk) | 4/4 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SFP Dialysate (N=4) | Standard Dialysate (N=7)
Chest Pain (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SFP Dialysate (N=4) | Standard Dialysate (N=7)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Air Embolism (Vascular disorders) | 0 (0) | 1 (1)
Arteriovenous Fistula Site Complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arteriovenous Fistula Thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Asthenia (General disorders) | 0 (0) | 1 (1)
Blindness (Eye disorders) | 1 (1) | 0 (0)
Blood Pressure Diastolic Increased (Investigations) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Breath Sounds Abnormal (Investigations) | 2 (2) | 2 (4)
Cardiac Murmur (Investigations) | 0 (0) | 1 (1)
Carotid Bruit (Investigations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 1 (1) | 1 (2)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Device Leakage (General disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (2)
Dizziness (Nervous system disorders) | 3 (13) | 3 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Eye Haemorrhage (Eye disorders) | 0 (0) | 2 (2)
Eyelid Oedema (Eye disorders) | 0 (0) | 1 (1)
Face Oedema (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Fluid Retention (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Flushing (Vascular disorders) | 1 (1) | 0 (0)
Gingival Infection (Infections and infestations) | 0 (0) | 1 (1)
Haemodialysis Complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Haemodialysis-induced Symptom (Injury, poisoning and procedural complications) | 2 (4) | 1 (2)
Headache (Nervous system disorders) | 1 (1) | 3 (4)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (2) | 2 (6)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 3 (9) | 1 (1)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 3 (3)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (3)
Neoplasm Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (7)
Peripheral Coldness (Vascular disorders) | 0 (0) | 1 (1)
Post-traumatic Pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural Hypertension (Injury, poisoning and procedural complications) | 2 (2) | 3 (7)
Procedural Hypotension (Injury, poisoning and procedural complications) | 3 (6) | 4 (8)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Rales (Respiratory, thoracic and mediastinal disorders) | 1 (8) | 3 (6)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Swelling (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 3 (7)
Thrombosis in Device (General disorders) | 1 (1) | 0 (0)
Traumatic Arthropathy (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Vascular Access Complication (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Vascular Graft Thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Visual Acuity Reduced (Eye disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (3)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Study suspended after 1st 11 subjects enrolled. Study design changed significantly upon re-initiation, so 1st 11 subjects analyzed for safety only; no efficacy. Efficacy analysis from study after re-initiation is found under protocol NIH-FP-01 PRIME.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes